CLINICAL TRIAL: NCT06692907
Title: A Phase 2b, Double-Blind, Placebo Controlled Trial to Evaluate the Efficacy of Intramuscularly Administered CssBA+dmLT Against Moderate-severe Diarrhea in a Controlled Human Infection Model With Enterotoxigenic Escherichia Coli (ETEC) Strain B7A in Healthy Adults
Brief Title: Efficacy Study of IM Administered CssBA+dmLT Against Moderate-severe Diarrhea in Human Infection Model With ETEC Strain B7A in Healthy Adults
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 23-0006; 5UM1AI148684-04 (NIH)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-07-18

CONDITIONS: Escherichia Infection
Keywords: B7A; Controlled; Diarrhea; Double-Blind; ETEC; Health Adult; IM Administered; Infection Model; Phase 2B; Vaccine
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Study staff including Outcomes Assessor, Study Statistician, Study Regulatory, QC coordinators and lab staff.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1A (Experimental): Participants will receive 45 mcg CssBA with 0.5 mcg dmLT vaccine intramuscular injection on Days 1, 22 and 43, outpatient. Participants who meet challenge criteria will orally receive 1x10^10 cfu of ETEC strain B7A, inpatient, approximately 28 days after the third dose of study agent. N= 18.
  Interventions: Other: B7A (ETEC challenge strain); Biological: CssBA; Biological: dmLT
- Cohort 1B (Placebo Comparator): Participants will receive 0.6 mL of 0.9% normal saline intramuscular injection on Days 1, 22 and 43, outpatient. Participants who meet challenge criteria will orally receive 1x10^10 cfu of ETEC strain B7A, inpatient, approximately 28 days after the third dose of study agent . N= 18.
  Interventions: Other: B7A (ETEC challenge strain); Other: Placebo
- Cohort 2A (Experimental): Participants will receive 45 mcg CssBA with 0.5 mcg dmLT vaccine intramuscular injection on Days 1, 22 and 43, outpatient. Participants who meet the challenge criteria will orally receive 1x10^10 cfu of ETEC strain B7A, inpatient, approximately 28 days after the third dose of study agent. N= 18.
  Interventions: Other: B7A (ETEC challenge strain); Biological: CssBA; Biological: dmLT
- Cohort 2B (Placebo Comparator): Participants will receive 0.6 mL of 0.9% normal saline intramuscular injection on Days 1, 22 and 43, outpatient. Participants who meet the challenge criteria will orally receive 1x10^10 cfu of ETEC strain B7A, inpatient, approximately 28 days after the third dose of study agent. N= 18.
  Interventions: Other: B7A (ETEC challenge strain); Other: Placebo

INTERVENTIONS:
Other: B7A (ETEC challenge strain) — A pathogenic strain of ETEC that can cause illness ranging from mild watery diarrhea to severe symptoms. The primary complication associated with an infection from this strain is dehydration.
Biological: CssBA — A CS6 based vaccine against ETEC (Enterotoxigenic Escherichia coli) in preventing moderate-severe diarrhea obtained via purification from a host E. coli expression strain, BL21(DE3), harboring a pET24a (+) plasmid containing the CssBA gene expressing the his-tagged CssBA protein.
  Arms: Cohort 1A; Cohort 2A
Biological: dmLT — An E. coli double mutant heat labile toxin. This genetically attenuated strain is expressed from a plasmid (pLC403) in the E. coli expression strain JM83.
  Arms: Cohort 1A; Cohort 2A
Other: Placebo — Placebo
  Arms: Cohort 1B; Cohort 2B

SUMMARY:
The study is designed to evaluate the safety, immunogenicity, and efficacy of the intramuscular administration of a CS6 based vaccine (CssBA) against ETEC co-administered with double mutant labile toxin (dmLT) in preventing moderate-severe diarrhea (MSD) following challenge with ETEC strain B7A in healthy adults. Approximately 72 adult participants, divided into 4 cohorts of 18, will be randomized 1:1 to receive vaccine (45 micrograms CssBA with 0.5 micrograms dmLT) or placebo (normal saline) on an outpatient basis. All participants will receive 3 intramuscular (IM) doses of vaccine or placebo at 3-week intervals (days 1, 22 and 43). Following vaccination, participants will be followed as outpatients for safety using a memory aid from the time of each vaccination through 7 days post each vaccination. Approximately 28 days (plus or minus 1 day) after receipt of the 3rd dose of study agent, participants meeting challenge criteria will be admitted to an inpatient unit and be administered an oral dose of 1 x 10^10 cfu (colony-forming unit) of ETEC strain B7A. Five days after challenge, participants will be treated with ciprofloxacin, except in cases of known allergy or intolerance. Participants will be discharged from the inpatient unit when they have completed their 3-day antibiotic course and are able to care for themselves. After discharge from the inpatient unit, participants will return for clinic visits and have a phone visit to provide any updates on medication, medical history and AE/SAEs. The primary objectives are: 1) Estimate CssBA+dmLT efficacy in preventing moderate-severe diarrhea (MSD) following challenge with ETEC strain B7A in healthy adults. 2) Evaluate the safety of intramuscular injection of CssBA+dmLT.

DETAILED DESCRIPTION:
The study is designed to evaluate the safety, immunogenicity, and efficacy of the intramuscular administration of a CS6 based vaccine (CssBA) against ETEC co-administered with double mutant labile toxin (dmLT) in preventing moderate-severe diarrhea (MSD) following challenge with ETEC strain B7A in healthy adults.

Approximately 72 adult participants, divided into 4 cohorts of 18, will be randomized 1:1 to receive vaccine (45 micrograms CssBA with 0.5 micrograms dmLT) or placebo (normal saline) on an outpatient basis. All participants will receive 3 intramuscular (IM) doses of vaccine or placebo at 3-week intervals (days 1, 22 and 43). Following vaccination, participants will be followed as outpatients for safety using a memory aid from the time of each vaccination through 7 days post each vaccination. Approximately 28 days (plus or minus 1 day) after receipt of the 3rd dose of study agent, participants meeting challenge criteria will be admitted to an inpatient unit and be administered an oral dose of 1 x 10^10 cfu (colony-forming unit) of ETEC strain B7A. After receipt of challenge agent, the participant will fast for 90 minutes. Participants will be monitored daily for diarrhea and other signs/symptoms of enteric illness. All stool will be collected and graded, and loose stools (grade 3-5) will be weighed. Five days after challenge (or earlier if clinically indicated), participants will be treated with ciprofloxacin, except in cases of known allergy or intolerance in which case trimethoprim-sulfamethoxazole will be used. Participants will be discharged from the inpatient unit when they have completed their 3-day antibiotic course and are able to care for themselves, including maintaining hydration status. Follow-up outpatient visits for 5 days and 4 weeks after discharge will monitor safety and immunologic parameters, and a phone visit will be conducted 6 months after last dose of study agent. The primary objectives are: 1) Estimate CssBA+dmLT efficacy in preventing moderate-severe diarrhea (MSD) following challenge with ETEC strain B7A in healthy adults. 2) Evaluate the safety of intramuscular injection of CssBA+dmLT. The secondary objectives are: 1)Determine illness severity following ETEC B7A challenge in participants who received CssBA+dmLT vs placebo using an evidence-based disease severity score (1). 2)Evaluate ETEC CS6- and LT-specific serum IgG and IgA responses following vaccination and challenge. 3)Evaluate ETEC CS6- and LT-specific IgG and IgA in Antibodies from Lymphocyte Supernatant (ALS) following vaccination and 4) Determine the prevalence and duration of fecal shedding of B7A following challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant, non-breast-feeding adults, age 18 to 49 years (inclusive) at the time of enrollment.
2. Willing and able to sign and date informed consent document prior to study procedures.
3. Stated willingness to be available for all study visits and comply with all trial procedures throughout the duration of the trial, including adherence to Lifestyle Considerations.
4. Participants of childbearing potential must have a negative pregnancy test at study enrollment.
5. For participants of childbearing potential*: agree to use highly effective contraception with heterosexual intercourse for at least 1 month prior to the first vaccination through at least two months after receipt of the challenge agent or last dose of study product if not challenged. True abstinence is also acceptable.

   * Childbearing potential in a participant assigned female at birth is defined as not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal.
   * Acceptable forms of highly effective contraception for participants assigned female at birth include same sex relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the participant enrollment, barrier methods such as condoms or diaphragms with spermicide, effective intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill"). Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.
6. Body mass index (BMI) 19 to less than 40 kg/m^2 at screening.
7. In good health. As determined by medical history and physical examination to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of safety of participants and interpretations of the scientific aims of the trial. Chronic medical diagnoses/conditions should be stable for the last 60 days (no hospitalizations, ER, or urgent care for condition or need for supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis/condition in the 60 days before enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or done for financial reasons, and in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the Principal or sub-Investigator licensed to make medical diagnosis, will not be considered a deviation of this inclusion criterion. Participants may be on chronic or as needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to participant safety or assessment of reactogenicity and immunogenicity, and do not indicate a worsening of medical diagnosis/condition. Similarly, medication changes subsequent to enrollment and trial vaccination are acceptable provided the change was not precipitated by deterioration in the chronic medical condition, and there is no anticipated additional risk to the participant or interference with the evaluation of responses to trial vaccination.
8. Oral temperature is less than 100.4 degrees Fahrenheit (38 degrees Celsius) at the time of enrollment.
9. Heart rate (HR) 60 to 100 beats per minute, inclusive. If participant baseline HR is between 50 and 60 beats per minute and the Principal or sub-Investigator licensed to make medical diagnosis determines that this is not clinically significant (e.g., if they are known to be high intensity athletes, have no clinical symptoms associated with the bradycardia, and have no signs or symptoms of other diseases causing bradycardia), this will NOT be considered a grade 1 adverse event and the participant still will be eligible.
10. Blood pressure (BP):systolic BP >/= 90 to </= 140 mm Hg; diastolic BP >/=55 to </=90 mmHg.
11. Must agree to refrain from donating blood or plasma (outside of this trial) from the first dose of study product until at least 30 days after completion of inpatient portion of the trial or last day of study product if not challenged.

Exclusion Criteria:

1. Abnormal stool pattern (fewer than 3 stools per week or more than 3 stools per day) on a regular basis; loose or liquid stools on other than an occasional basis.
2. History of microbiologically confirmed ETEC or cholera infection in the last 3 years.
3. Symptoms consistent with MSD concurrent with travel to countries where ETEC infection is endemic (refer to MOP section for a list of endemic countries) within 3 years prior to enrollment.
4. Vaccination for, ingestion of or occupational handling of ETEC, cholera, or E. coli heat labile toxin within 3 years prior to enrollment.
5. Any condition that, in the judgment of the investigator, precludes participation because it could affect participant safety or endpoint evaluation.
6. Unable to understand spoken and written English.
7. Venous access deemed inadequate for phlebotomy/cannulation needs of the study.
8. Have any disease or medical condition that, in the opinion of the Principal or sub-Investigator licensed to make medical diagnosis, is a contraindication to study participation. These include:

   * History within the past 12 months of inflammatory bowel disease (IBD) (including ulcerative colitis, Crohn's disease, indeterminate colitis, or celiac disease), irritable bowel syndrome (IBS), or any active uncontrolled gastrointestinal disorders or diseases as assessed by the investigator.
   * Within the past 12 months have symptoms or evidence of active gastritis or severe gastroesophageal reflux disease not well controlled on medication, gastric surgery, or gastric acid hyper-secretory disorders (e.g., Zollinger-Ellison syndrome), gastrointestinal obstruction, ileus, gastric retention, bowel perforation, toxic colitis, persistent infectious gastroenteritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection.
9. Known active neoplastic disease (non-melanoma, treated, skin cancers are permitted), a history of any hematologic malignancy, or have used anticancer chemotherapy/radiation therapy (cytotoxic) within 3 years prior to study enrollment.
10. Positive serology results for HIV Ag/Ab combo, HBsAg, or HCV Ab.
11. Serum IgA <40 mg/dL
12. History of immunodeficiency due to congenital or hereditary causes, underlying illness, or treatment
13. Have screening labs that are greater than Grade 1 severity. Values below the lower limit of normal for creatinine, bilirubin and/or ALT are acceptable for study inclusion as they are not considered to be clinically significant by the Principal or sub-Investigator licensed to make medical diagnosis.
14. Within the past 3 years have participated in an ETEC challenge study or reports having received vaccination for ETEC.
15. Use of immunosuppressive/immunomodulating disease therapy within 1 year of 1st dose of study vaccine.
16. Planning to receive Ig or other blood products (with exception of Rho D Ig) from 90 days before 1st vaccination until 30 days after receipt of challenge agent or last day of study product if not challenged.
17. Received systemic antibiotics* within 7 days prior to receipt of study vaccine.

    *Including Quinolones, nitrofurantoin, nalidixic acid, chloramphenicol, Quinine, chloroquine, primaquine.
18. Took prescription or OTC medication containing loperamide, acetaminophen, aspirin, ibuprofen, or other non-steroidal anti-inflammatory within 24 hours of receipt of vaccine.
19. Planning to receive an investigational agent or product* within 30 days prior to the first study vaccination through 60 days after last dose of study vaccine.

    *Including vaccine, drug, biologic, device, blood product, or medication, other than from participation in this trial.
20. Planning to receive a licensed, live vaccine within 30 days before or after each vaccination.
21. Planning to receive a licensed, inactivated vaccine* within 14 days before or after each vaccination: *An exception is a COVID and/or influenza vaccine which may be received within 7 days of vaccination and still be eligible.
22. Within 14 days prior to vaccination, have completed a course of oral or parenteral* corticosteroids of any dose for 5 or more days, or high dose** inhaled corticosteroids.

    * Including intra-articular

    **High dose defined per guideline; https://www.nhlbi.nih.gov/files/docs/guidelines/asthma_qrg.pdf
23. Known hypersensitivity to both ciprofloxacin and trimethoprim-sulfamethoxazole; sodium bicarbonate; or any components of vaccine, placebo, or challenge material.
24. Have a history of severe reactions following previous immunization with any licensed or unlicensed vaccine.
25. Have a history of alcohol or drug abuse within 1 year prior to enrollment.
26. Positive urine toxicology screen for opiates
27. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 3 years prior to enrollment.
28. Taking or have taken prescription or over-the-counter medication for weight reduction 3 months before enrollment through the completion of the challenge phase.
29. Within 7 days after discharge from the challenge unit plan to work in either a patient care setting, day care center, or as a food handler.
30. Plan to have daily contact with individuals with possible increased susceptibility* to severe ETEC infection* in the week after discharge from the inpatient challenge unit.

    * Increased susceptibility to severe ETEC infection including; Immunocompromised elderly persons aged 70 years or more, diapered individuals, persons with disabilities, children <2 years old, a woman known to be pregnant or nursing, or anyone with diminished immunity. Known daily contact includes contact at home, school, day-care, nursing home, or similar places.
31. History of prolonged QT syndrome and/or torsade de pointes or in those with risk factors for QT syndrome, such as currently receiving Class IA or Class III antiarrhythmic agents, tricyclic antidepressants, or antipsychotics.
32. Currently known to have a folate deficiency, or a history of glucose-6-phosphate dehydrogenase deficiency.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of CssBA+dmLT injected participants experiencing local solicited AEs | Through 7 days after vaccination
Number and percentage of CssBA+dmLT injected participants experiencing MAAEs | Through 6 months after last vaccination
Number and percentage of CssBA+dmLT injected participants experiencing SAEs | Through 6 months after last vaccination
Number and percentage of CssBA+dmLT injected participants experiencing systemic solicited AEs | Through 7 days after vaccination
Number and percentage of CssBA+dmLT injected participants experiencing unsolicited AEs | Through Day 71
Number and percentage of participants experiencing moderate-severe diarrhea (MSD) with Enterotoxigenic Escherichia coli (ETEC) | Day 70-79
  MSD is defined as experiencing >/=4 loose/liquid stools or >/= 400 g of loose/liquid stools in any 24-hour period during inpatient stay.

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) summarizing the maximum observed antigen-specific CS6 IgG antibody titers by Antibodies from Lymphocyte Supernatant (ALS) | Day 8 - Day 99
GMT of summarizing maximum observed antigen-specific dmLT IgG antibody titer by ALS | Day 8 -Day 99
GMT summarizing maximum observed antigen-specific dmLT IgA antibody titer by ALS | Day 8 -Day 99
GMT summarizing the maximum observed antigen-specific CS6 IgA antibody titers by ALS | Day 8 - Day 99
Mean severity of ETEC B7A-associated diarrhea | Day 70 - Day 79
  ETEC B7A disease severity score calculated from three components that are evaluated daily during the ETEC Challenge. ETEC B7A disease severity scores will only be calculated for participants who receive a dose of ETEC B7A.
Median number of days with a positive stool culture for B7A following challenge | Day 70 - Day 79
Number and percentage of participants with >/= 4-fold rise from baseline in antigen-specific CS6 antibody titer to IgA in serum | Through Day 99
Number and percentage of participants with >/= 4-fold rise from baseline in antigen-specific CS6 antibody titer to IgG in serum | Through Day 99
Number and percentage of participants with >/= 4-fold rise from baseline in antigen-specific dmLT antibody titer to IgA in serum | Through Day 99
Number and percentage of participants with >/= 4-fold rise from baseline in antigen-specific dmLT antibody titer to IgG in serum | Through Day 99
Number and percentage of participants with a positive stool culture for B7A | Day 71 - Day 79

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio